CLINICAL TRIAL: NCT02338271
Title: Safety and Efficacy Study of Autologous Adipose Derived Mesenchymal Stem Cells Implantation in Chronic Low Back Pain Patients With Lumbar Intervertebral Disc Degeneration
Brief Title: Autologous Adipose Derived Stem Cell Therapy for Intervertebral Disc Degeneration
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inbo Han (Other)
Collaborators: CHA University (Other)
Responsible Party: Sponsor-Investigator, Inbo Han, Associate Professor, Spine Neurosurgeon, Bundang CHA Hospital
Organization: Bundang CHA Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADMSC-DD-Han
Record Dates: First submitted 2015-01-07; First posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Low Back Pain
Keywords: Low back pain; Mesenchymal stromal stem cell; Hyaluronic acid
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- a single, open clinical trial (Other): a single-group, open, investigator-initiated clinical study
  : autologous adipose derived mesenchymal stem cell (2 x 10^7 cells/mL /vial or 4 x 10^7 cells/mL /vial) plus Tissuefill (hyaluronic acid derivatives) 1mL/syringe
  Interventions: Other: autologous adipose derived mesenchymal stem cell

INTERVENTIONS:
Other: autologous adipose derived mesenchymal stem cell — autologous adipose derived mesenchymal stem cell (2 x 10^7 cells/mL /vial or 4 x 10^7 cells/mL /vial) and Tissuefill (hyaluronic acid derivatives) 1mL/syringe

SUMMARY:
1. Subject: 10 patients

   : Chronic low back pain patients with lumbar intervertebral disc degeneration
2. Investigational Product

   : Autologous adipose derived mesenchymal stem cells plus hyaluronic acid derivatives (Tissuefill)
3. Time frame

   * 1 year

DETAILED DESCRIPTION:
1. Purpose of the Clinical Study

   : To transplant autologous adipose derived mesenchymal stem cells with hyaluronic acid to patients with chronic low back pain caused by a degenerative lumbar disc to examine the procedure's safety and efficacy.
2. Phases and Design of the Clinical Study

   : This clinical study is a I/IIa phase single-group, open, investigator initiated trial.
3. Investigational Product : Autologous adipose derived mesenchymal stem cells separated from the subject (2 x 10^7 cells/mL /vial or 4 x 10^7 cells/mL /vial).

The investigational product mixed with 1 mL of the concomitant drug Tissuefill (hyaluronic acid derivatives, Cha Meditech Co., Ltd.).

4. Inclusion Criteria

1. Males and female subjects aged 18 or over and less than 70.
2. Subjects who have experienced pain in the lower back or buttocks who have failed to respond to conservative therapies performed for a period of 3 months or longer.
3. Oswestry Disability Index of 30 % or higher.
4. Visual Analogue Scale of 4 or higher.
5. Subjects who have received a Magnetic Resonance Imaging (hereinafter referred to as MRI) assessment of grades 3 to 4 for Lumbar 1 - Sacral 1, according to the Pfirrmann grading system.
6. Subjects who are assessed to have a similar degree of pain as usual when a discogram is performed on the degenerative lumbar disc(s) identified by MRI, having one or two discs that cause the concordant pain.
7. Subjects who have signed the informed consent form for stem cell transplantation therapy.

5. Exclusion Criteria

1. Subjects with severe lumbar stenosis or herniated nucleus pulposus in the lumbar exhibiting symptoms of nerve compression and requiring surgery.
2. Subjects with spinal instability, spondylitis, or vertebral fractures
3. Patients with severe intervertebral disc degeneration that has resulted in a reduction of the disc height by ½ or more.
4. Subjects with severe osteoporosis (with an average T-score of -2.5 or below in the lumbar bone density test)
5. Patients who have received intra-discal procedures such as stem cell therapy or the injection of steroids into the disc or surgery such as discectomy on the disc on which the cell transplantation is planned to be performed.
6. Patients who have received a lumbar epidural steroid injection within a week prior to the cells transplantation.
7. Subjects who are hypersensitive to sodium hyaluronate.
8. Pregnant or breastfeeding women
9. Female patients with the possibility of pregnancy during the period of the clinical study who are not using a medically acceptable method of contraception.
10. Subjects with mental illness or a drug or alcohol addiction or subjects who are incapable of understanding the purpose and method of this clinical study.
11. Subjects who have participated in another clinical study in the 30 days prior to this study.
12. Subjects with a severe medical disease (hypertension unresponsive to drug treatment, diabetes unresponsive to drug treatment, hepatocirrhosis, renal failure, tumor) that can affect the outcome of this clinical study.
13. Subjects with any other clinically significant findings that renders the subject unsuitable for the clinical study, as judged by the investigator responsible for the clinical study.

6. Dosage and Administration

: The autologous adipose derived mesenchymal stem cell as the investigational product (2 x 10^7 cells/mL /vial or 4 x 10^7 cells/mL /vial) and Tissuefill 1mL/syringe are supplied to the operating room. The investigational product and the Tissuefill (hyaluronic acid derivatives) are mixed and placed in a 22 G syringe. A single dosage of 2ⅹ10^7 autologous adipose derived mesenchymal stem cells per person is administered on 5 subjects, and a single dosage of 4ⅹ10^7 cells per person is administered on 5 subjects, injected into the center of the nucleus pulposus.

7. Primary Endpoint: Evaluation of Safety and Tolerability The transplantation will be considered to be safe and tolerable, in the absence of the following types of counterevidence.

- Adverse events of grade 3 (NCI grading system) or above related to the cell products/ any evidence that the cells were contaminated by pollutants / any evidence that the cells exhibit tumorigenic potential

8. Secondary Endpoint

1. Change in the T2 MRI signal intensity of the nucleus pulposus in autologous adipose derived mesenchymal stem cells at 6 and 12 months after the transplantation compared to before the transplantation
2. Change in the VAS at 1, 3, 6, 9, and 12 months after the transplantation of autologous adipose derived mesenchymal stem cells, compared to before the transplantation
3. Change in the ODI at 1, 3, 6, 9, and 12 months after the transplantation of autologous adipose derived mesenchymal stem cells, compared to before the transplantation
4. Change in the Short Form (SF)-36 at 1, 3, 6, 9, and 12 months after the transplantation of autologous adipose derived mesenchymal stem cells, compared to before the transplantation
5. Assessment of the overall improvement in the Disc Height Index (hereinafter referred to as DHI) at 6 and 12 months after the transplantation of autologous adipose derived mesenchymal stem cells, compared to before the transplantation

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have experienced pain in the lower back or buttocks who have failed to respond to conservative therapies performed for a period of 3 months or longer.
2. Oswestry Disability Index of 30% or higher.
3. Visual Analogue Scale of 4 or higher.
4. Subjects who have received a Magnetic Resonance Imaging (hereinafter referred to as MRI) assessment of grades 3 to 4 for Lumbar 1 - Sacral 1, according to the Pfirrmann grading system.
5. Subjects who are assessed to have a similar degree of pain as usual when a discogram is performed on the degenerative lumbar disc(s) identified by MRI, having one or two discs that cause the pain.
6. Subjects who have signed the informed consent form for stem cell transplantation therapy.

Exclusion Criteria:

1. Subjects with severe lumbar stenosis or herniated nucleus pulposus in the lumbar exhibiting symptoms of nerve compression and requiring surgery.
2. Subjects with spinal instability, spondylitis, or vertebral fractures
3. Patients with severe intervertebral disc degeneration that has resulted in a reduction of the disc height by ½ or more.
4. Subjects with severe osteoporosis (with an average T-score of -2.5 or below in the lumbar bone density test)
5. Patients who have received intra-discal procedures such as stem cell therapy or the injection of steroids into the disc or surgery such as discectomy on the disc on which the cell transplantation is planned to be performed.
6. Patients who have received a lumbar epidural steroid injection within a week prior to the cells transplantation.
7. Subjects who are hypersensitive to sodium hyaluronate.
8. Pregnant or breastfeeding women
9. Female patients with the possibility of pregnancy during the period of the clinical study who are not using a medically acceptable method of contraception.

   * Medically acceptable methods of contraception: condoms, an oral contraceptive administered continually for at least 3 months, an implantable contraceptive surgically inserted 3 months prior to the clinical study, injected or inserted contraceptives, an intrauterine contraceptive device, etc.
10. Subjects with mental illness or a drug or alcohol addiction or subjects who are incapable of understanding the purpose and method of this clinical study.
11. Subjects who have participated in another clinical study in the 30 days prior to this study.
12. Subjects with a severe medical disease (hypertension unresponsive to drug treatment, diabetes unresponsive to drug treatment, hepatocirrhosis, renal failure, tumor) that can affect the outcome of this clinical study.
13. Subjects with any other clinically significant findings that renders the subject unsuitable for the clinical study, as judged by the investigator responsible for the clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Safety and Tolerability (Adverse events) | 12months
  The transplantation will be considered to be safe and tolerable, in the absence of the following types of counter evidence.
  - Adverse events of grade 3 (NCI grading system) or above related to the cell products/ any evidence that the cells were contaminated by pollutants / any evidence that the cells exhibit tumorigenic potential.
  Adverse events will be reported at 1, 3, 6, 9, and 12 months

SECONDARY OUTCOMES:
Change in the T2 MRI signal intensity of the nucleus pulposus | 12months
  Change in the T2 MRI signal intensity of the nucleus pulposus in autologous adipose derived mesenchymal stem cells at 6 and 12 months after the transplantation compared to before the transplantation
Overall improvement in the Disc Height Index | 12months
  Assessment of the overall improvement in the Disc Height Index at 6 and 12 months after the transplantation of autologous adipose derived mesenchymal stem cells, compared to before the transplantation
improvement in Visual Analogue Scale (VAS) | 12 months
  Change in the VAS at 1, 3, 6, 9, and 12 months after the transplantation of autologous adipose derived mesenchymal stem cells, compared to before the transplantation
improvement in Oswestry Disability Index (ODI) | 12 months
  Change in the ODI at 1, 3, 6, 9, and 12 months after the transplantation of autologous adipose derived mesenchymal stem cells, compared to before the transplantation
improvement in Short Form-36 | 12 months
  Change in the Short Form (SF)-36 at 1, 3, 6, 9, and 12 months after the transplantation of autologous adipose derived mesenchymal stem cells, compared to before the transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Inbo Han, MD, PhD, Principal Investigator — CHA Bundang Medical Center
Locations (1):
- CHA University, CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kumar H, Ha DH, Lee EJ, Park JH, Shim JH, Ahn TK, Kim KT, Ropper AE, Sohn S, Kim CH, Thakor DK, Lee SH, Han IB. Safety and tolerability of intradiscal implantation of combined autologous adipose-derived mesenchymal stem cells and hyaluronic acid in patients with chronic discogenic low back pain: 1-year follow-up of a phase I study. Stem Cell Res Ther. 2017 Nov 15;8(1):262. doi: 10.1186/s13287-017-0710-3. PMID 29141662